CLINICAL TRIAL: NCT06721221
Title: Impact of Catheter Stability on the Outcomes With Very High Power Short Duration Ablation
Acronym: SVtag
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM/8942-1/2023; BWI-IIS-688 (Other Grant/Funding Number: Biosense Webster)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation Ablation; Pulmonary Vein Isolation
Keywords: pulmonary vein isolation; catheter stability; first-pass isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SVtag arm. Point-by-point PVI with the Svtag software (Experimental): PVI will be performed with QDot Micro catheter in QMODE plus with the Svtag software.
  Interventions: Device: Point-by-point PVI with the QDot Micro catheter in QMODE+ setting with the Svtag software

INTERVENTIONS:
Device: Point-by-point PVI with the QDot Micro catheter in QMODE+ setting with the Svtag software — PVI will be performed via femoral access after transseptal puncture, guided by fluoroscopy pressure monitoring, intracardiac echocardiography (ICE) or transesophageal echocardiography (TEE). A fast anatomical left atrial map will be created; then, point-by-point PVI will be performed with QDot Micro catheter in QMODE plus with the Svtag software. Inter-tag distance should be ≤ 6 mm on the posterior wall and ≤ 4 mm on the anterior wall. All applications' duration should be 4 seconds. After creating the isolation circle, the presence or absence of first-pass isolation will be assessed on each side by the presence of entrance block. If PVI is complete, this is defined as first-pass isolation. If PVI is not complete at this point, touch-up lesions will be delivered to reach the isolation of all pulmonary veins. After that, acute PV reconnections will be evaluated during a 20 minutes waiting period.

SUMMARY:
Background: Atrial fibrillation (AF), the most common cardiac rhythm disorder can be treated with pulmonary vein isolation (PVI). One technique for PVI is point-by-point radiofrequency ablation. Very high power short duration ablation is one of the most advanced technologies for radiofrequency ablation. However, acute efficacy results with this technology vary in a wide range. Improvements in automated tagging modules, incorporating tracking of cardiac and respiratory motion and enhanced stability algorithms, may allow for a better assessment of lesion quality and location and may improve the so called first-pass isolation rate (an indicator for acute procedural efficacy).

Objective: To assess the acute procedural outcomes of very high power short duration PVI with the new enhanced stability software.

Methods: Investigator-initiated, prospective, single-arm study on one hundred symptomatic patients with paroxysmal AF will undergo PVI with the QDOT catheter using a power setting of 90W(QMODE+). The inter-tag distance will be 6 mm posteriorly and 4 mm anteriorly, and the enhanced stability algorithm will be used in all cases. After creating the isolation circle, the presence or absence of first-pass isolation will be assessed on each side by the presence of entrance block. Primary endpoint will be first-pass isolation rate. Secondary outcomes are as follows: procedure time, left atrial dwell time, RF time, number of RF tags, use of a steerable sheath, occurrence of serious adverse events.

Hypothesis: Very high power short duration PVI using the new stability software results in a higher rate of first-pass isolation than previously published.

DETAILED DESCRIPTION:
Background Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia in adults. Its prevalence increases with age, affecting 3/100 people, and its incidence is also correlated with age, affecting 30/100.000 people per year. Its clinical significance stems from common complications (stroke, heart failure) and concomitant higher mortality. The most effective rhythm control treatment method for atrial fibrillation is catheter ablation, which seeks to maintain sinus rhythm. Isolation of the triggering pulmonary veins (PVI) from the left atrium is the cornerstone of AF ablation. PVI has undergone significant technical development over the past decade; however, the chances of arrhythmia recurrence and the occurrence of procedural complications are not negligible. Experiments have shown that lesions with a slightly smaller surface diameter and less depth develop during high power short duration (HPSD) ablation. The shorter ablation time might result in more consistent lesion creation if the catheter stability is good during the radiofrequency (RF) application. On the other hand, if the catheter position is unstable during the RF application, a huge variety might occur between the created lesion sizes. Regarding the safety aspects, the shallower lesions might cause less damage to the surrounding tissues. The latest application of HPSD technology is the so-called "very high power short duration" (vHPSD) ablation with application of 90W power for 3-4 seconds. The ablation index does not work for such a short ablation time; thus, other lesion-predicting parameters should be used, such as impedance drop and catheter stability. At the moment, there are two software products for ablation point visualization. The commercially available legacy software was originally built to assess catheter stability over a long ablation period (e.g. with the ablation index), but the system is unable to differentiate between poor and good catheter stability during a 4 seconds time frame. Conversely, the new SVTAG software is adapted to assess catheter stability over a 4-second period; thus, the operator might get better feedback on the actual lesion creation. This might result in a more optimized lesion set and a more effective PVI, but this hypothesis has not been tested yet.

Objective: To evaluate the acute efficacy of radiofrequency PVI performed with 90W, using the new stability software version.

Primary hypothesis: Pulmonary vein isolation is effective with the Svtag software that gives proper feedback on catheter stability, resulting in short procedures, high first-pass isolation rate, and few acute reconnections.

Study Design: Multicenter, prospective, single-arm study.

Research period: The planned research period starts in the first quarter of 2023 until December 2025.

Study subjects: Planned number of included subjects: 150. Inclusion criteria: Symptomatic paroxysmal or persistent AF, Age >18 years, Willingness to sign the informed consent form.

Exclusion criteria: Contraindication to ablation, Contraindication of long-term anticoagulation, Long-standing persistent AF, History of PVI, History of cardiac surgery, Pregnancy, Active malignancy, Life expectancy <1 year, Valvular AF, Reversible cause of AF (e.g. hyperthyroidism).

Study procedure: PVI will be performed via femoral access after transseptal puncture, guided by fluoroscopy pressure monitoring, intracardiac echocardiography (ICE) or transesophageal echocardiography (TEE). A fast anatomical left atrial map will be created; then, point-by- point PVI will be performed with QDot Micro catheter in QMODE plus with the Svtag software. Inter-tag distance should be ≤ 6 mm on the posterior wall and ≤ 4 mm on the anterior wall. All applications' duration should be 4 seconds. After creating the isolation circle, the presence or absence of first-pass isolation will be assessed on each side by the presence of entrance block. If PVI is complete, this is defined as first-pass isolation. If PVI is not complete at this point, touch-up lesions will be delivered to reach the isolation of all pulmonary veins. After that, acute PV reconnections will be evaluated during a 20 minutes waiting period. In case of acute reconnection, additional applications will be delivered to complete the PVI. No further waiting is necessary after that.

Primary endpoint: First-pass isolation rate.Secondary endpoints: Occurrence of any adverse events related to the procedure during the hospital stay and 1 month after the procedure. Acute reconnection: pulmonary vein reconnection during the 20 minutes waiting period. Impact of scar burden in the on the FPI rate assessed by EA mapping (during the waiting period). 12-month AF-free survival

Nature of the study: Investigator-initiated clinical trial, there is no commissioning company. The study is not for commercial gain. Not a drug test. Subjects will not undergo any additional procedures in connection to the study. The study protocol is in compliance with routine clinical practice, no additional radiation is applied.

Adverse events: PVI is a routinely used, safe procedure these days. During the current clinical trial, for the participating patients, there is no additional intervention that is different from the everyday routine, except for the 20-minute waiting period after the PVI. During the procedure, patients are exposed to the following potential complications, which in total occur in 1% of cases: Complications involving the vascular access site: femoral pseudoaneurysm / arterio- venous fistula / hematoma with bleeding requiring blood transfusion, Pericardial fluid, Pericardial tamponade, Stroke / TIA, Esophageal injury / perforation / fistula, Myocardial infarction, Phrenic nerve paresis, Pulmonary vein stenosis, Conduction system damage requiring pacemaker implantation, Death. The participating centers' Electrophysiology Laboratories are prepared and capable of providing fast and adequate care for these complications.

Statistical analysis: Continuous variables are expressed as means and standard deviations, or medians and interquartile ranges, depending on the normal or non-normal distribution. Categorical variables are expressed in numbers and percentages. Continuous variables are compared by parametric or non-parametric tests, depending on the distribution, while categorical variables are compared by Chi-square test or Fisher's exact test. A two-tailed p-value of <0.05 is considered statistically significant. Statistical analyses will be performed using IBM SPSS 25 (Apache Software Foundation, USA) and GraphPad Prism 7.1 (GraphPad Softwares Inc., USA) software, or other statistical software products.

Data management: All study patient data is entered into an electronic database (REDCap) in a coded and unique manner, with a unique identifier, to which project staff has a password-protected, defined level of access. Each person involved in the study is given a unique identification code, and the data stored in the database is linked to that unique identifier. Thus, a data set will be incomprehensible and unusable for an external (unauthorized) user. The data belonging to the unique identification code, with which the patient's identity can be clearly indicated (name, place and date of birth, clinical reference number, identification number, identity card number, etc.) are not available from the database and are stored separately from it. Access to personal data will be limited to authorized staff (both clinical and research) at the local hospital site.

Funding: A research grant is provided by the Johnson and Johnson Company.

Ethics approval: An ethics approval application is submitted separately in case of all participating centers to their national or local ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal or persistent AF
* Age >18 years
* Willingness to sign the informed consent form

Exclusion Criteria:

* Contraindication to ablation
* Contraindication of long-term anticoagulation
* Long-standing persistent AF
* History of PVI
* History of cardiac surgery
* Pregnancy
* Active malignancy
* Life expectancy <1 year
* Valvular AF
* Reversible cause of AF (e.g. hyperthyroidism).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
First-pass isolation rate | Endpoint is assessed intra-procedurally
  After creating the isolation circle, the presence or absence of first-pass isolation will be assessed on each side by the presence of entrance block. If PVI is complete, this is defined as first-pass isolation. If PVI is not complete at this point, touch-up lesions will be delivered to reach the isolation of all pulmonary veins.

SECONDARY OUTCOMES:
Acute reconnection | Assessed 20 minutes after PVI is reached during the procedure
  Pulmonary vein reconnection during the 20 minutes waiting period
12-months AF freedom | 12-month from procedure
  Freedom from AF during 12-month follow-up
Complications or adverse events | 1 month
  Occurrence of any adverse events related to the procedure during the hospital stay and 1 month after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Heart and Vascular Center, Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
All study patient data is entered into an electronic database (REDCap) in a coded and unique manner, with a unique identifier, to which project staff has a password-protected, defined level of access. Each person involved in the study is given a unique identification code, and the data stored in the database is linked to that unique identifier. Thus, a data set will be incomprehensible and unusable for an external (unauthorized) user. The data belonging to the unique identification code, with which the patient's identity can be clearly indicated (name, place and date of birth, clinical reference number, identification number, identity card number, etc.) are not available from the database and are stored separately from it. Access to personal data will be limited to authorized staff (both clinical and research) at the local hospital site.

REFERENCES:
- [Background] Reddy VY, Grimaldi M, De Potter T, Vijgen JM, Bulava A, Duytschaever MF, Martinek M, Natale A, Knecht S, Neuzil P, Purerfellner H. Pulmonary Vein Isolation With Very High Power, Short Duration, Temperature-Controlled Lesions: The QDOT-FAST Trial. JACC Clin Electrophysiol. 2019 Jul;5(7):778-786. doi: 10.1016/j.jacep.2019.04.009. Epub 2019 May 8. PMID 31320006
- [Background] Kewcharoen J, Techorueangwiwat C, Kanitsoraphan C, Leesutipornchai T, Akoum N, Bunch TJ, Navaravong L. High-power short duration and low-power long duration in atrial fibrillation ablation: A meta-analysis. J Cardiovasc Electrophysiol. 2021 Jan;32(1):71-82. doi: 10.1111/jce.14806. Epub 2020 Nov 18. PMID 33155303
- [Background] Nakagawa H, Ikeda A, Sharma T, Govari A, Ashton J, Maffre J, Lifshitz A, Fuimaono K, Yokoyama K, Wittkampf FHM, Jackman WM. Comparison of In Vivo Tissue Temperature Profile and Lesion Geometry for Radiofrequency Ablation With High Power-Short Duration and Moderate Power-Moderate Duration: Effects of Thermal Latency and Contact Force on Lesion Formation. Circ Arrhythm Electrophysiol. 2021 Jul;14(7):e009899. doi: 10.1161/CIRCEP.121.009899. Epub 2021 Jun 17. PMID 34138641
- [Background] Hussein A, Das M, Riva S, Morgan M, Ronayne C, Sahni A, Shaw M, Todd D, Hall M, Modi S, Natale A, Dello Russo A, Snowdon R, Gupta D. Use of Ablation Index-Guided Ablation Results in High Rates of Durable Pulmonary Vein Isolation and Freedom From Arrhythmia in Persistent Atrial Fibrillation Patients: The PRAISE Study Results. Circ Arrhythm Electrophysiol. 2018 Sep;11(9):e006576. doi: 10.1161/CIRCEP.118.006576. PMID 30354288
- [Background] Taghji P, El Haddad M, Phlips T, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Evaluation of a Strategy Aiming to Enclose the Pulmonary Veins With Contiguous and Optimized Radiofrequency Lesions in Paroxysmal Atrial Fibrillation: A Pilot Study. JACC Clin Electrophysiol. 2018 Jan;4(1):99-108. doi: 10.1016/j.jacep.2017.06.023. Epub 2017 Sep 27. PMID 29600792
- [Background] Solimene F, Schillaci V, Shopova G, Urraro F, Arestia A, Iuliano A, Maresca F, Agresta A, La Rocca V, De Simone A, Stabile G. Safety and efficacy of atrial fibrillation ablation guided by Ablation Index module. J Interv Card Electrophysiol. 2019 Jan;54(1):9-15. doi: 10.1007/s10840-018-0420-5. Epub 2018 Jul 30. PMID 30058055
- [Background] Szegedi N, Sallo Z, Perge P, Piros K, Nagy VK, Osztheimer I, Merkely B, Geller L. The role of local impedance drop in the acute lesion efficacy during pulmonary vein isolation performed with a new contact force sensing catheter-A pilot study. PLoS One. 2021 Sep 16;16(9):e0257050. doi: 10.1371/journal.pone.0257050. eCollection 2021. PMID 34529678
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505